CLINICAL TRIAL: NCT00963534
Title: Lenalidomide, Bendamustine and Rituximab as First-line Therapy for Patients Over 65 Years With Mantle Cell Lymphoma - a Nordic Lymphoma Group Trial
Brief Title: Lenalidomide, Bendamustine and Rituximab as First-line Therapy for Patients Over 65 Years With Mantle Cell Lymphoma.
Acronym: LENA-BERIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Mundipharma Pte Ltd. (Industry); Celgene (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-MCL4
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Lenalidomide; Bendamustine; Rituximab; Nordic Lymphoma Group; MTD for lenalidomide; Untreated patients; Patients with mantle cell lymphoma, age over 65 years
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lenalidomide, bendamustine, rituximab (Experimental)
  Interventions: Drug: lenalidomide, bendamustine, rituximab

INTERVENTIONS:
Drug: lenalidomide, bendamustine, rituximab — Phase I: Maximally tolerable dose of lenalidomide will be determined, starting with 5 mg per day, and up to maximally 25 mg per day. This treatment is given in combination with bendamustine and rituximab.
  Phase II: Determination of progression free survival with treatment with lenalidomide (dosing determined in phase I) in combination with bendamustine and rituximab.
Drug: lenalidomide, bendamustine, rituximab — lenalidomide: day 1-21, maximum 13 cycles bendamustine: days 1-2, cycle 1-6 rituximab: day1, cycle 1-6

SUMMARY:
In phase I: Establishing maximally tolerated dose of lenalidomide in combination with bendamustine and rituximab.

In phase II: Evaluation of progression free survival with treatment with lenalidomide, bendamustine and rituximab

DETAILED DESCRIPTION:
This trial consists of both a phase I portion and a phase II portion. In phase I, the MTD of lenalidomide is determined, starting with 5 mg/day given up to maximally 25 mg/day. In combination with this treatment, bendamustine and rituximab are given at fixed doses.

The phase I portion follows a sequential dose escalation, 3+3 design. Initially, three subjects are started treatment with dose regimen 1 (5 mg/day). After the third subject completed two cycles of treatment, if no DLT has occured, the next group of three subjects are treated at the next dose level of lenalidomide (10 mg/day). If one of the three initial subjects experiences a DLT, the cohort is expanded to six subjects. If less than two out of the six subjects experiences a DLT, then the next higher dose group is initiated. If two or more subjects experiences a DLT, no higher dose levels will be tested and the MTD dose has been exceeded.

Additional subjects are enrolled at the MTD on the phase II portion of the trial.

The above described treatment with lenalidomide, bendamustine and rituximab are given in 6 cycles, cycle length 22 days. Lenalidomide is given day 1-21, bendamustine day 1-2 and rituximab day 1. During the following maintenance treatment, single treatment with lenalidomide will be given with the same dose of lenalidomide (25 mg/day) for 7 cycles, whether in phase I or phase II portion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years, or age under 65 years, unable to tolerate high dose chemotherapy with autologous stem cell support
* Histologically confirmed mantle cell lymphoma, stage II-IV at time of diagnosis
* No previous treatment for lymphoma except radiotherapy or one cycle of any chemotherapy regimen for lymphoma
* WHO Performance Status 0-3
* Written informed concent
* Female subjects of childbearing potential must agree to use and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, through study drug therapy and for 4 weeks after the end of study drug therapy
* Male subjects must agree to use condoms throughout study drug therapy if their partner is of childbearing potential, and has no contraception, and agree to not donate semen during study drug therapy and for one week after end of study drug therapy
* All subjects must agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation, and agree not to share study medication with another person

Exclusion Criteria:

* Impaired liver function
* ANC less than 1.0 x 10 9, unless caused by bone marrow infiltration by lymphoma
* Platelet count less than 60 x 10 9, unless caused by bone marrow infiltration by lymphoma
* Creatinine clearance below 50 ml/min (cockcroft formula))
* Known HIV positivity
* Known seropositivity for HCV, HBsAG, anti-HBc, or other active infection uncontrolled by treatment
* Psychiatric illness or condition which could interfere with the subject´s ability to understand the requirements of the study
* Requirement of corticosteroid therapy at a dose over 10 mg prednisolone/day
* Pregnant or lactating females

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide (phase I) Progression free survival (phase II) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jerkeman, MD, PhD, Principal Investigator — University Hospital Lund, Sweden; Jan Sundberg, RN, Study Director — University Hospital Lund, Sweden
Locations (17):
- Denmark (3):
  - Århus University Hospital, Aarhus
  - Herlev Hospital, Copenhagen
  - Rigshospitalet, Department of Hematology, Copenhagen
- Helsinki University Central Hospital, Helsinki, Finland
- Norway (5):
  - Haukeland University Hospital, Department of Oncology, Bergen
  - Norwegian Radium Hospital, Oslo
  - Ulleval University Hospital, Department of Oncology, Oslo
  - University Hospital of Stavanger, Department of Haematology and Oncology, Stavanger
  - University Hospital of Tromso, Department of Oncology, Tromsø
- Sweden (8):
  - Sahlgrenska University Hospital, Department of Hematology, Gothenburg
  - University Hospital Linköping, Department of Hematology, Linköping
  - Sunderbyn Hospital, Department of Medicine, Luleå
  - University Hospital Lund, Department of Oncology, Lund
  - Karolinska University Hospital, Department of Hematology, Stockholm
  - Sundsvall Hospital, Department of Medicine, Sundsvall
  - University Hospital of Norrland, Department of Oncology, Umeå
  - Uppsala University Hospital, Department of Oncology, Uppsala

REFERENCES:
- [Derived] Albertsson-Lindblad A, Kolstad A, Laurell A, Raty R, Gronbaek K, Sundberg J, Pedersen LB, Ralfkiaer E, Karjalainen-Lindsberg ML, Sundstrom C, Ehinger M, Geisler C, Jerkeman M. Lenalidomide-bendamustine-rituximab in patients older than 65 years with untreated mantle cell lymphoma. Blood. 2016 Oct 6;128(14):1814-1820. doi: 10.1182/blood-2016-03-704023. Epub 2016 Jun 27. PMID 27354719